CLINICAL TRIAL: NCT03790943
Title: Prospective Single Center Cohort Study for Early Detection of Cardiac Dysfunction in Childhood Cancer Survivors
Brief Title: Cardiac Dysfunction in Childhood Cancer Survivors
Acronym: Cardio-Onco
Status: Recruiting | Type: Observational
Sponsor: University of Bern (Other)
Collaborators: University Hospital, Basel, Switzerland (Other); University Children's Hospital Basel (Other); Insel Gruppe AG, University Hospital Bern (Other); Cantonal Hospital of St. Gallen (Other); Luzerner Kantonsspital (Other); University Hospital, Geneva (Other)
Responsible Party: Sponsor
Other Study IDs: SCCSS_cardiac_FU
Record Dates: First submitted 2018-06-25; First posted 2019-01-02 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Dysfunction; Cardiovascular Diseases; Childhood Cancer
Keywords: Childhood cancer survivors; Late effects; Cardiotoxicity; Chemotherapy; Anthracyclines; Radiation
MeSH Terms: conditions — Cardiovascular Diseases; Neoplasms; Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: cardiac assessment — Personal history, physical examination including anthropometry with hip/waist-ratio, electrocardiogram, echocardiography, 1-minute-sit-to-stand test, questionnaires on health-related quality of life (SF-36), diet, physical activity, and fatigue

SUMMARY:
This multicenter, prospective cohort study evaluates early cardiac dysfunction in adult survivors of childhood cancer. The hypothesis of this study is that cardiac dysfunction can be detected earlier when using speckle tracking echocardiography as novel echocardiographic technique compared to conventional echocardiography.

DETAILED DESCRIPTION:
Cardiovascular disease including cardiac dysfunction is the leading non-malignant cause of death in childhood cancer survivors. Early detection of cardiac dysfunction is important to identify those in need for medical intervention to improve outcome. This study invites adult childhood cancer survivors to a clinical appointment to the University Hospital Bern, Switzerland. A detailed, standardized cardiac assessment including conventional and novel echocardiographic techniques (speckle tracking) as well as cardiopulmonary exercise testing is performed. Cardiac dysfunction is evaluated in survivors who have had cardiotoxic cancer therapy with anthracyclines and/or chest radiation (high risk) and in survivors who have had chemotherapy other than anthracyclines (standard risk).

ELIGIBILITY:
This prospective cohort study is nested within the Childhood Cancer Registry (ChCR), a national, population-based cancer registry that includes all children and adolescents in Switzerland who were diagnosed with cancer at age 0-20 years. It includes patients diagnosed with leukemia, lymphoma, central nervous system tumors, and malignant solid tumours or Langerhans cell histiocytosis. Childhood cancer survivors have survived at least 5 years from cancer diagnosis.

Inclusion Criteria:

* Registered in the ChCR
* Formerly treated at the Department of Pediatric Hematology/Oncology of one of five participating centers
* Treated with any chemotherapy and/or chest radiation
* Survived ≥ 5 years since most recent cancer diagnosis (primary cancer, relapse(s), secondary cancer) at time of examination
* Diagnosed at age ≤ 20 years
* ≥ 18 years of age at time of study participation
* Resident in Switzerland
* Written informed consent

Exclusion Criteria:

* Study participants will be excluded if they do not meet the above mentioned inclusion criteria or refuse to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult survivors of childhood cancer, formerly treated at the University Children's Hospital Bern or University Children's Hospital Basel or Children's Hospital of Eastern Switzerland or Children´s Hospital Lucerne or University Hospitals of Geneva, with any chemotherapy and/or chest radiation.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-02-13 (Actual); Primary Completion 2029-04-23 (Estimated); Study Completion 2029-04-23 (Estimated)

PRIMARY OUTCOMES:
Prevalence of cardiac dysfunction | Baseline and longitudinal follow-up where clinically indicated
  Conventional echocardiography: left ventricular ejection fraction (%)
Prevalence of cardiac dysfunction | Baseline and longitudinal follow-up where clinically indicated
  Speckle tracking echocardiography: longitudinal (LS), circumferential (CS), and radial strain (RS)
Prevalence of impaired exercise capacity | Baseline
  Cardiopulmonary exercise testing: peak oxygen consumption, percent-predicted carbon dioxide production
Treatment-related risk factors | Baseline
  Cumulative doses of anthracyclines, steroids, and alkylating agents (mg/m2)
Treatment-related risk factors | Baseline
  Dose of chest radiation (Gray)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia E Kuehni, MD, Principal Investigator — University of Bern
Locations (6):
- Switzerland (6):
  - Department of Cardiology, University Hospital Basel, Basel, Canton of Basel-City
  - Institute of Social and Preventive Medicine, University of Bern, Bern, Canton of Bern
  - Department of Cardiology, Inselspital Bern, Bern
  - Department of Cardiology, University Hospitals of Geneva, Geneva
  - Department of Cardiology, Lucerne Cantonal Hospital, Lucerne
  - Department of Cardiology, Cantonal Hospital of St. Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schindera C, Kuehni CE, Pavlovic M, Haegler-Laube ES, Rhyner D, Waespe N, Roessler J, Suter T, von der Weid NX. Diagnosing Preclinical Cardiac Dysfunction in Swiss Childhood Cancer Survivors: Protocol for a Single-Center Cohort Study. JMIR Res Protoc. 2020 Jun 10;9(6):e17724. doi: 10.2196/17724. PMID 32269016